CLINICAL TRIAL: NCT05800067
Title: A Single-arm Prospective Trial of Axicabtagene Ciloleucel (Axi-cel) Retreatment in Relapsed/Refractory Large B-cell Lymphoma
Brief Title: Axi-cel Retreatment in Relapsed/Refractory LBCL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FKC876-LBCL-001
Record Dates: First submitted 2022-12-02; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2022-08

CONDITIONS: CAR-T Retreatment
Keywords: Axi-cel retreatment, R/R LBCL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Axi-cel (Experimental): Patients will receive a target dose of 2×10⁶ Axi-cel per kilogram of body weight after receiving a conditioning regimen. The conditioning regimen and dosage will be at investigator's discretion based on patient's status.
  Interventions: Drug: axi-cel

INTERVENTIONS:
Drug: axi-cel — Axicabtagene ciloleucel (Axi-cel) is an autologous anti-CD-19 chimeric antigen receptor(CAR) T-cell therapy approved by FDA in 2017 for the treatment of patients with relapsed/refractory large B-cell lymphoma (R/R LBCL). Now, it is the standard treatment for these patients recommended by NCCN and other guidelines. Axi-cel was approved for R/R LBCL patients who had received 2 or more prior lines of therapy on 2021 June in China.

SUMMARY:
This is a prospective, single-arm, clinical study to explore the efficacy and safety of Axi-cel retreatment in R/R LBCL in Shanghai Ruijin Hospital in China.

R/R LBCL patients who treated with Axi-cel got non-CR or relapsed were eligible for Axi-cel retreatment in this study. Patients will receive the standard dose of Axi-cel and follow the standard process. Other related treatment like bridging therapy or combination therapy will be based on patients status and investigators' decision. The primary endpoint is ORR, the secondary endpoint is CR, PR, DOR, PFS, OS and AE. A total of 32 patients is planned to be enrolled in this study. The trial will not go on if nobody got CR or PR in first 6 patients.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open-label two-stage study. There were 6 cases enrolled in Phase 1 and 26 cases enrolled in Phase 2, for a total of 32 cases.

This study aimed to collect data on efficacy and safety after secondary infusion treatment with aquilencel in adult patients with r/r LBCL after the first treatment of CD19 CAR-T. No form of grouping was performed in this study, and subgroup analyses were performed based on the actual data collected.

Research Process:

The patient has been evaluated for disease after the first treatment of akilencel, and the investigator decided to give the patient a second treatment based on clinical practice. Obtain informed consent before the second treatment of CD19 CAR-T, collect data on the patient's disease status before the second dose, previous and current decontamination treatment and other related treatments, and perform imaging tests such as positron emission tomography and computed tomography (PET-CT) or electronic computed tomography (CT) on the same day, day 15, day 29, month 3 after secondary administration, and 6, 9, 12, 18 and 24 months after secondary administration to confirm the collection of efficacy data, and investigators evaluated data on adverse events related to CD19 CAR-T, related laboratory results, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent Form (ICF);
2. Adults with diagnosed relapsed or refractory Large B-cell lymphoma who have completed initial treatment with Axi-cel;
3. non-CR or relapsed after the initial Axi-cel infusion;
4. CD19 status by lymphoma lesion biopsy is at the discretion of investigators.
5. Antidrug antibodies (ADA) of Axi-cel should be performed prior to retreatment. 6) Lymphodepleting chemotherapy (fludarabine and cyclophosphamid) related toxicities were ≤ grade 1 or at the base line of Axi-cel initial treatment.

8）No serious adverse events occurred during the initial Axi-cel treatment or the adverse events in the first treatment period have recovered.

Exclusion Criteria:

1. Patients with hypersensitivity to any active ingredient or excipients (dimethyl sulfoxide, compound electrolyte injection, human albumin);
2. Uncontrolled systemic fungal, bacterial, viral, or other infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-03-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Best objective response rate | Up to 2 years
  ORR, defined as the incidence of either a complete response or a partial response assessed by investigators according to Lugano 2014 criteria.

SECONDARY OUTCOMES:
Complete response (CR) rate | Up to 2 years
  Complete response assessed by investigators according to Lugano 2014 criteria.
Duration of Response (DOR) | Up to 2 years
  Among subjects who experience an objective response, DOR is defined as the date of their first objective response (which is subsequently confirmed) to disease progression per the revised IWG Response Criteria for Malignant Lymphoma or death regardless of cause. Subjects not meeting the criteria for progression or death by the analysis data cutoff date will be censored at their last evaluable disease assessment date and their response will be noted as ongoing.
Progression-Free Survival (PFS) | Up to 2 years
  PFS is defined as the time from the axicabtagene ciloleucel infusion date to the date of disease progression per the revised IWG Response Criteria for Malignant Lymphoma or death from any cause. Subjects not meeting the criteria for progression by the analysis data cutoff date will be censored at their last evaluable disease assessment date.
Overall Survival (OS) | Up to 2 years
  OS is defined as the time from axicabtagene ciloleucel infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at their last contact date.

CONTACTS AND LOCATIONS:
Overall Officials: weili Zhao, MD,PhD, Study Chair — Ruijin hospital,China
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No